CLINICAL TRIAL: NCT05878366
Title: Understanding and Maximizing the Community Impact of Antimalarial Treatment (INDIE-SMC)
Acronym: INDIE-SMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Groupe de Recherche Action en Sante (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 29193; INV-053846 (Other Grant/Funding Number: BMGF)
Record Dates: First submitted 2023-05-09; First posted 2023-05-26 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2024-01

CONDITIONS: Malaria; Malaria,Falciparum
Keywords: Plasmodium falciparum; Seasonal Malaria Chemoprevention; Antimalarial treatment; Burkina Faso; SP+AQ
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Intervention Model Description: This study involves and Operational evaluation of a modified existing intervention delivered in independent clusters. The project and its implementation are prepared in direct interaction with the Ministry of Health (MoH) to tailor data collection to local needs.
Masking Description: Laboratory analysis and impact analysis teams will be blinded to intervention arm.
  Entomology staff involved in the mosquito feeding assays will be blinded for the parasitology results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Active Comparator): SMC in children under the age of 5 years, implemented by the MoH without directly observed treatment for the full course of SMC
  Interventions: Other: Seasonal Malaria Chemoprophylaxis (under 5 year old) implemented by the MoH without DOT
- Arm 2 (Experimental): SMC in children under the age of 5 years, with directly observed treatment for the full course of SMC
  Interventions: Other: Seasonal Malaria Chemoprophylaxis (under 5 years old) with DOT
- Arm 3 (Experimental): SMC in children under the age of 10 years, with directly observed treatment for the full course of SMC
  Interventions: Other: Seasonal Malaria Chemoprophylaxis (under 10 years old) with DOT

INTERVENTIONS:
Other: Seasonal Malaria Chemoprophylaxis (under 5 year old) implemented by the MoH without DOT — Standard approach for SMC strategy used by the Ministry of Health (without directly-observed therapy) and without any interference of the study team. Implemented over 4 rounds, carried out in June-October 2023 with ~30 days between rounds.
  Arms: Arm 1
Other: Seasonal Malaria Chemoprophylaxis (under 5 years old) with DOT — SMC will be implemented with the same number of rounds and the same timing as in active comparator arm but village health workers will visit the participants at home to administer each dose of study treatment (with DOT-directly-observed therapy)
  Arms: Arm 2
Other: Seasonal Malaria Chemoprophylaxis (under 10 years old) with DOT — SMC will be implemented as in arm 2 but age of participants is extended up to 10 years: each dose of study treatment (with DOT-directly-observed therapy) distributed at home by village health workers.
  Arms: Arm 3

SUMMARY:
Seasonal Malaria Chemoprophylaxis (SMC) is a fundamental component of malaria control. The SMC program involves that sulfadoxine-pyrimethamine plus amodiaquine (SPAQ) is given to children below the age of 5 years during the peak transmission season in areas of seasonal malaria transmission. Yet, its efficacy is increasingly below expectations.

This study involves an Operational evaluation of a modified existing intervention and its implementation are prepared in direct interaction with the Ministry of Health (MoH) to tailor data collection to local needs. The main questions it aims to answer are:

1. what are the reasons for the continued high infection rates in the SMC-targeted population;
2. what are the implications for transmission of sub-optimal SMC in children less than 5 years old;
3. can the impact of SMC be improved by including older age groups that would both expand the population that experiences direct chemoprophylactic benefits and concurrently reduce transmission to the wider community

Researchers will:

i) Compare SMC effectiveness as implemented by the national malaria control program and SMC implemented in a research context where all doses are directly observed.

ii) Quantify the infectious reservoir and the contribution of different age groups to transmission with conventional SMC (<5 years) and extended SMC (<10 years) iii) Determine the impact of drug resistance and drug absorption on SMC efficacy iv) Understand social barriers and enablers interfering with SMC efficacy and how SMC uptake is related to health equity with special attention to gender inequalities.

v) Quantify SMC efficacy decay under programmatic conditions and key drivers of this decay.

DETAILED DESCRIPTION:
Seasonal Malaria Chemoprophylaxis is a well established method of malaria control. Sulfadoxine-pyrimethamine plus amodiaquine (SPAQ) is given to children below the age of 5 years during the peak transmission season in areas of seasonal malaria transmission. Whilst highly effective in controlled research studies, the impact of SMC in terms of reducing infection prevalence is less following operational delivery. It is currently unclear why and what drivers of SMC coverage and uptake play a role. In addition, the relative importance of parasite drug resistance, limited adherence, poor drug absorption and frequent re-infections remain largely unexplored.

Lastly, the World Health Organization has recently widened the scope for SMC to target all vulnerable populations. The Ministry of Health (MoH) in Burkina Faso is considering extending SMC to all children below 10 years of age; the impact of SMC on clinical incidence and parasite prevalence in this population with markedly different immunity is unknown. Moreover, this older age group is known to be highly relevant for onward malaria transmission, making it important to quantify the impact of SMC on the human infectious reservoir for malaria and broader benefits to the community.

The investigators propose a cluster-randomized trial in Saponé Health District, Burkina Faso, with three study arms:

i. SMC in children under the age of 5 years, implemented by the MoH without directly observed treatment for the full course of SMC ii. SMC in children under the age of 5 years, with directly observed treatment for the full course of SMC iii. SMC in children under the age of 10 years, with directly observed treatment for the full course of SMC The investigators will deliver the different arms of the intervention to 40 clusters of 3 households/compounds (i.e. 120 compounds per arm). The primary endpoint is parasite prevalence at the end of the malaria transmission season, secondary endpoints include the impact of SMC on clinical incidence, gametocyte carriage and potential for onward parasite transmission to mosquitoes. As relevant factors in determining these efficacies, drivers of SMC uptake and treatment adherence will be determined, as well as drug concentrations, parasite resistance markers and transmission of parasites to mosquitoes.

ELIGIBILITY:
The study population will be derived from individuals aged 3 months to up to 10 years old eligible for SMC.

Inclusion criteria:

* Eligible for chemoprevention for SMC as per the current recommendations
* Age 3- 59 months for arms i. and ii.
* Age 60 months up to 10 years old for arm iii.
* Absence of symptomatic falciparum malaria, defined by fever on enrolment
* Absence of other non-P. falciparum species on blood film
* No evidence of acute severe or chronic disease
* Able and willing to comply with the study protocol and follow-up schedule
* Parent or guardian provides written, informed consent on behalf of child

Exclusion criteria:

* Symptoms of malaria (axillary fever ≥ 37.5 °C and/or history of fever in the past 48 hours)
* Previous reaction to study drugs / known allergy to study drugs
* Signs of severe malaria, including hyperparasitemia (defined as asexual parasitemia > 100,000 parasites / µL)
* Signs of acute or chronic illness, including hepatitis
* The use of other medication (except for paracetamol and/or aspirin)
* Presence of severe malnutrition according to WHO's child growth standards

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2978 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Parasite prevalence by quantitative PCR (qPCR) at the end of the transmission season in age groups targeted by seasonal malaria chemoprevention. | 4 weeks
  This endpoint will be compared between arms 1 and 2 (in children aged 3-59 months) and arms 2 and arm 3 (in children aged 3 months-9 years).

SECONDARY OUTCOMES:
Parasite prevalence by microscopy at the end of the transmission season in all age groups | 4 weeks
  This endpoint will compare the parasite prevalence in all age groups between intervention arms.
Parasite prevalence by qPCR at the end of the transmission season in all age groups | 4 weeks
  This endpoint will compare the parasite prevalence in all age groups between intervention arms.
Parasite prevalence by microscopy prior to SMC rounds 2, 3 and 4 in SMC-targeted age groups | 8 weeks
  This endpoint will compare the prevalence by microscopy before SMC rounds (2, 3 and 4) between intervention arms.
Rate of re-infection with P. falciparum at weeks 3, 4 and 5 after the last round of SMC, assessed in SMC-targeted age groups | 10 weeks
  This endpoint will assess the rate of malaria reinfection at different time points after the alst round of SMC between intervention arms
Gametocyte prevalence by qRT-PCR at weeks 3, 4 and 5 after the last round of SMC, assessed in SMC-targeted age groups | 10 weeks
  This endpoint will compare the gametocyte prevalence between intervention arms at different time points after the last round of SMC.
Gametocyte prevalence by qRT-PCR at the end of the transmission season in all age groups | 8 weeks
  This endpoint will compare the gametocyte prevalence between intervention arms in all age groups
Plasma levels of AQ and DESAQ after the 4th round of SMC in children aged 3 months-9 years | 6 weeks
  This endpoint will compare the plasma levels of AQ and DESAQ between intervention arms.
Clinical malaria incidence captured during passive-case detection (between arm comparison) | Across study period (6 months)
  This endpoint will compare the cases of malaria between intervention arms.
Parasite prevalence by qPCR at the end of the transmission season compared between arms 1 and combined arms 2 + 3. | 4 weeks
  This endpoint will assess the prevalence in targeted age groups in combined arms with similar treatment and population
Gametocyte prevalence by qRT-PCR at the end of the transmission season in age groups targeted by SMC (comparison between arm1 and 2 (in children aged 3-59 months) and arms 2 and arm 3 (in children aged 5 years-9 years). | 4 weeks
  This endpoint will assess the gametocyte prevalence and the end of the study between groups and combined similar groups.

OTHER OUTCOMES:
Infectivity to mosquitoes, defined as the percentage of infected mosquitoes, in relation to gametocyte density and plasma drug levels of AQ and DESAQ | Up to 10 weeks
  This endpoint will assess the infectivity to mosquitoes between intervention arms related to gametocytemia and plasma drug levels.
Size and age-distribution of the infectious reservoir for malaria | Through study completion, an average of 10 months
  This endpoint will assess the likelihood that a mosquito becomes infected with malaria parasites after feeding on a population member (between arm comparison)
Prevalence of drug resistance markers in infected children aged 3 months-9 years assessed post each round of SMC (between arm comparison) | Through study completion, an average of 10 months
  This endpoint will assess the prevalence of drug resistance markers after each round of SMC.
Description of perceived social barriers to SMC uptake | Through study completion, an average of 10 months
  This endpoint is designed to understand potential factors that influence SMC uptake and effectiveness
Quantification of SMC efficacy decay under programmatic conditions | Through study completion, an average of 10 months
  This endpoint will assess the practical realities that result in reduction of SMC coverage.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Tiono, PhD, MD, Principal Investigator — Groupe de Recherche Action en Sante
Locations (1):
- Groupe de Recherche Action en Santé, Ouagadougou, Burkina Faso

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised individual participant data may be shared on a digital repository or upon reasonable request.

REFERENCES:
- [Derived] Moreno M, Barry A, Gmeiner M, Yaro JB, Serme SS, Byrne I, Ramjith J, Ouedraogo A, Soulama I, Grignard L, Soremekun S, Koele S, Ter Heine R, Ouedraogo AZ, Sawadogo J, Sanogo E, Ouedraogo IN, Hien D, Sirima SB, Bradley J, Bousema T, Drakeley C, Tiono AB. Understanding and maximising the community impact of seasonal malaria chemoprevention in Burkina Faso (INDIE-SMC): study protocol for a cluster randomised evaluation trial. BMJ Open. 2024 Mar 12;14(3):e081682. doi: 10.1136/bmjopen-2023-081682. PMID 38479748

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT05878366/SAP_000.pdf